CLINICAL TRIAL: NCT04922307
Title: Reduction of Allogenic Blood Transfusion in Locally Advanced Kidney Cancer
Acronym: RESTRICT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kelvin Moses, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#202548
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Kidney Cancer
Keywords: nephrectomy; blood sparing; allogenic blood transfusion
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Sparing Protocol (Experimental): The intervention group (120 patients) will undergo radical nephrectomy with blood-sparing techniques. Acute Normovolemic Hemodilution (ANH) collects patients own blood prior to the start of surgical procedure; Cell saver is the collection of blood lost during surgery with subsequent auto-transfusion of the patients own cells; Veno-venous bypass will be used for patients with anticipated large loss of blood during surgery (>1L). The patients in the interventional group will be blinded to which blood sparing techniques utilized.
  Interventions: Procedure: Blood Sparing Protocol
- Standard Blood Replacement (Active Comparator): The control group of one hundred and twenty (120) patients will undergo radical nephrectomy without blood sparing techniques (ie. Standard of care). Patients who need blood transfusion will receive cross-matched allogenic blood products.
  Interventions: Procedure: Standard Blood Replacement

INTERVENTIONS:
Procedure: Blood Sparing Protocol — Acute Normovolemic Hemodilution, Cell Saver, and/or Veno-venous Bypass
  Arms: Blood Sparing Protocol
Procedure: Standard Blood Replacement — Allogenic blood transfusion as determined intra-operatively
  Arms: Standard Blood Replacement

SUMMARY:
The Reduction of Allogenic Blood Transfusion in Locally Advanced Kidney Cancer Trial (RESTRICT).

The primary objective is to reduce the number of units of allogenic blood transfusion in locally advanced kidney cancer (≥ cT2). Secondary objectives include reduction in perioperative complications, assessment of recurrence free-survival and improving overall survival.

DETAILED DESCRIPTION:
The Reduction of Allogenic Blood Transfusion in Locally Advanced Kidney Cancer Trial (RESTRICT) is a randomized study to investigate blood sparing using autologous normovolemic hemodilution (ANH) or cell salvage at the time of nephrectomy for locally advanced kidney cancer after assessing inclusion criteria patients will be randomized to undergo standard blood management including the possibility of allogenic transfusion vs autologous blood transfusion. There are multiple ways patients can receive allogenic or autologous blood, including veno-venous bypass or cardiopulmonary bypass (typically reserved for patients with a thrombus above the level of the hepatic veins or entering the heart).

ELIGIBILITY:
Inclusion Criteria:

* Renal masses ≥ cT2 (by any conventional imaging).
* N1 or M1 disease is allowed if they are deemed surgical candidates (including cytoreductive nephrectomy).
* Male and female patients.
* 18 and older.
* Ejection fraction (EF) ≥ 45% by echocardiogram (ECHO).
* Adequate organ function as defined by:

  * Hemoglobin ≥ 9 g/dL. Pre-operative allogenic blood transfusion is allowed.
  * Platelets ≥ 100.000/μl.
  * Albumin ≥ 2.5 g/dL.
  * Aspartate Aminotransferase (AST) and alanine transaminase (ALT) ≤ 75U/L or total bilirubin ≤ 2.0 mg/dL.
  * WBC within institutional normal limits.
  * PT within institutional normal limits.
  * INR < 1.5 and PTT normal.
  * Consent and compliance with all aspects of the study protocol.

Exclusion Criteria:

* Male and female younger than 18 years old.
* Non-surgical candidate
* Unstable angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of units of allogenic blood transfusions | Baseline to 30 days postoperatively
  The primary goal of the study is to evaluate the impact of the blood sparing techniques on the reduction of allogenic blood transfusion in locally advanced kidney cancer. The total number of allogenic blood units used at the end of each case will be assessed

SECONDARY OUTCOMES:
Number of Complications | Baseline to 30 days and 90 days postoperatively
  Number of complications will be assessed by Clavien-Dindo Index
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions
  Grade II Pharmacological treatment with drugs other than such allowed for grade I.
  Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Not under general anesthesia
  * IIIb Under general anesthesia
  Grade IV Life-threatening complication (including CNS complications)* requiring IC/ICU- management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgan dysfunction
  Grade V Death
Grade of Complications | Baseline to 30 days and 90 days postoperatively
  Grade of complications will be assessed by Clavien-Dindo Index
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions
  Grade II Pharmacological treatment with drugs other than such allowed for grade I.
  Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Not under general anesthesia
  * IIIb Under general anesthesia
  Grade IV Life-threatening complication (including CNS complications)* requiring IC/ICU- management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgan dysfunction
  Grade V Death
Kidney Cancer Recurrence | Up to 3 years postoperatively
  Assessment of recurrence of kidney cancer by radiographic imaging (CT or MRI)
Overall Survival | Up to 3 years postoperatively
  Assessment of survival after surgery
Quality of life as measured by Functional Assessment of Cancer Therapy-Kidney Symptom Index (FSKI-19) | Pre-operative, 1 and 3 months postoperatively
  Assessment of quality of life measures postoperatively, scores range from 0-76, with higher scores indicating worse symptoms
  Score range: 0-76 A score of "0" is a severely symptomatic patient and the highest possible score is an asymptomatic patient.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Moses, Principal Investigator — Associate Professor
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No